CLINICAL TRIAL: NCT01800409
Title: Abdominal Functional Electrical Stimulation Training and Its Effect on Mechanical Insufflation-Exsufflation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GN12NE539
Record Dates: First submitted 2013-02-14; First posted 2013-02-27 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Cervical Spinal Cord Injury
Keywords: Tetraplegia
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFES training (Experimental): Participants will take part in AFES training sessions five times per week (Mon-Fri) for a total of 8 weeks During these sessions participants will receive AFES for 40 minutes. Training sessions are designed to strengthen the participants abdominal muscles in order to improve respiratory function
  Interventions: Device: AFES
- Control period (No Intervention): Four week control period. The order of the control and training periods will be randomised for each participant.

INTERVENTIONS:
Device: AFES — During the stimulation sessions electrical stimulation will be applied for 40 minutes per day, 5 days per week for a total of 8 weeks
  Other Names: neuromuscular stimulator (RehaStim, HasoMed, Germany)
  Arms: AFES training

SUMMARY:
Compromised respiratory function as a result of tetraplegia is a leading cause of rehospitalisation for the tetraplegic patient group. Electrical stimulation of the abdominal muscles has previously been used to improve the respiratory function of tetraplegic patients in the chronic stage of injury. In this study the investigators aim to evaluate the optimum protocol for the use of electrical stimulation of the abdominal muscles to improve the respiratory function of the tetraplegic population. The investigators also aim to investigate whether abdominal functional electrical stimulation combined with mechanical insufflation-exsufflation can be used to help further improve the respiratory function of the tetraplegic population.

DETAILED DESCRIPTION:
Respiratory infections are a leading cause of morbidity and mortality for the tetraplegic population. They are often caused by the build up of secretions in the lungs as a result of being unable to generate an effective cough. This inability to cough leads to many tetraplegic people requiring some type of intervention to aid the removal of secretions. Manually assisted coughing or routine suctioning through the patient's tracheostomy tube are commonly used. Both of these techniques are associated with problems: (i) Tracheostomy suctioning is uncomfortable and often misses the left bronchus, one of the contributing factors to 80% of pneumonia occurring in the left lung of the spinal cord injured population. (ii) A manually assisted cough is a safe and effective procedure but needs to be provided by a trained care giver with associated resource implications for the local health care provider. An alternative method to help clear secretions and improve ventilation is Mechanical Insufflation-Exsufflation (MI-E) where a combination of positive and negative pressure is applied to the user's airway in order to induce a cough. A number of studies have shown that MI-E is more effective at removing secretions and reducing respiratory infections than conventional suctioning and manually assisted cough techniques, with the advantage that secretions are removed from both bronchi. MI-E has also been shown to significantly reduce the length of ICU stay and reduce the rates of reintubation.

Individuals with tetraplegia have reduced exhaled tidal volume (VT) and reduced Cough Peak Flow (CPF) (maximum air flow rate during a cough. The CPF value can be used to assess the risk of respiratory infection, with a CPF < 160 L/min associated with no functional cough and a high risk of infection and a CPF of <270 L/min suggesting that a person will not be able to adequately clear secretions from their airway. The use of MI-E is therefore suggested for anyone with a CPF of <270 L/min.

Functional Electrical Stimulation (FES) is a technique which can be used to make paralysed muscles contract. The most effective contraction is observed when train of electrical pulses are applied close to the motor point of a paralysed muscle. When FES is applied to the abdominal muscles it is called Abdominal Functional Electrical Stimulation (AFES). AFES has previously been used to increase the VT and CPF of tetraplegic patients in a number of studies.

MI-E is routinely combined with manually assisted coughing in order to loosen lung secretions and to increase the user's CPF. In the same way as a manually assisted cough, AFES leads to increased abdominal movement, resulting in larger CPF. During recent studies the investigators have observed that the use of AFES with acute tetraplegic patients appears to be associated with an increased need for secretion clearance, indicating that AFES aids the loosening of lung secretions. Although the abdominal movement achieved with AFES is typically significantly smaller than that achieved with a manually assisted cough, it may have beneficial effects in combination with MI-E. In addition, AFES has the advantage that it can be applied consistently and requires less involvement of the caregiver.

The investigators hypothesise that (i) maximal respiratory improvements due to an AFES training programme will be achieved after more than 3 weeks of training, and (ii) that the combined use of AFES with MI-E may improve the respiratory function and ability to clear secretions of tetraplegic patients, resulting in a reduction in the number of respiratory infections in this group.

Methods

Participants Ten tetraplegic participants will be recruited for this study. All participants will be inpatients at the Queen Elizabeth National Spinal Injuries Unit, Southern General Hospital, Glasgow.

Experimental Procedures Each participant will undergo a pre study assessment. The study will take the form of a random crossover design involving a four week control period and an eight week training period which will be followed by a two week follow up period. The order of the control and training periods will be randomised for each participant. If the training period precedes the control period the follow up period will serve as a two week wash out period to avoid any carryover of acute effects from the training intervention. At the pre study assessment, and at the end of every second week, the participant will take part in an assessment session.

Pre study assessment Before the study commences each participant will undergo a pre study assessment which will also serve as a familiarisation session. Stimulation will be applied to the participant's abdominal muscles to test whether they respond to electrical stimulation. The optimum stimulation parameters (electrode position/frequency/current and pulsewidth) required to induce a strong contraction of the abdominal muscles will then be established. These stimulation parameters will be used as a starting point for the following training and assessment sessions. An assessment session, as outlined below, will then be conducted at the end of the pre study assessment.

Training sessions Participants will take part in AFES training sessions five times per week (Monday-Friday) for a total of 8 weeks. During these sessions participants will receive AFES for 40 minutes.

Assessment sessions Each participant will take part in bi-weekly assessment sessions throughout the study. At each assessment session a series of Forced Vital Capacity (FVC) tests will be performed with and without abdominal stimulation, which provide a measure of the participant's Vital Capacity (VC), Forced Exhaled Volume in one second (FEV1) and Peak Expiratory Flow (PEF). Respiratory flow and volume will be measured using a spirometer. To perform the FVC manoeuver the participant will be asked to inhale to Total Lung Capacity (TLC) and then exhale as quickly and as fully as they can. This will be repeated for each condition up to a maximum of 5 times, or until 3 attempts within 0.15L of each other are recorded. Many of the participants on this study will have a FVC of <1L. The ATS/ERS standards for spirometry suggest that for an FVC of <1L the range of acceptable values should be plus or minus 0.1L. All participants will perform the assessment sitting in an upright position.

The participant's cough peak flow (CPF) will also be measured under three conditions: (i) unassisted (ii) unassisted mechanical insufflation-exsufflation (MI-E) and (iii) MI-E assisted with Abdominal Functional Electrical Stimulation (AFES). To measure the CPF, five cycles of MI-E will be applied for both MI-E conditions. The maximum CPF value recorded from five attempts will be taken as the participant's CPF in each condition.

During the pre study assessment and at the end of the training and the control period an extended assessment session will be performed. The additional measurements will be (i) MI-E with manually assisted cough, and (ii) ultrasound measurement of diaphragm movement with and without AFES.

The CPF achieved using MI-E with a manually assisted cough will be recorded while the manually assisted cough is applied by the patient's regular caregiver, with the same caregiver applying the manually assisted cough in all three sessions.

The movement of the diaphragm will be measured during a FVC manoeuvre using an ultrasound probe, with and without AFES assistance. This will allow an evaluation of the effect of AFES on diaphragm movement.

Follow up/ Wash out period After the training period the participant will undergo a two week follow up period. If the participant has still to complete the control period this follow up will also act as a wash out. During this wash out period the participant will undergo no training sessions. The aim of this wash out period is to minimise the effect of any acute response from the training period to the control period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 16 years of age
* Reduced respiratory function as a result of a cervical spinal cord injury
* Good visual response to surface abdominal stimulation, suggesting that lower motor neurons are intact
* Ventilator independent

Exclusion Criteria:

* Under 16 years of age
* Female subjects who are pregnant
* Significant history of autonomic dysreflexia
* No visual response to surface abdominal stimulation, suggesting that lower motor neurons are not intact
* Unstable chest or abdominal injury
* High levels of intrinsic PEEP (bulleous disease, lung tumour etc)
* High anastomosis (e.g. oesophago-gastrectomy)
* Bulbar dysfunction
* Unable to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Respiratory function | at end of 8 week AFES intervention
  Forced Vital Capacity (FVC) tests will be performed with and without abdominal stimulation, which provides a measure of the participant's Vital Capacity (VC), Forced Exhaled Volume in one second (FEV1) and Peak Expiratory Flow (PEF). Respiratory flow and volume will be measured using a spirometer.

SECONDARY OUTCOMES:
the total excursion of the diaphragm under both stimulated and unstimulated conditions | at end of 8 week AFES intervention
  The movement of the diaphragm will be measured during a FVC manoeuvre using an ultrasound probe, with and without AFES assistance.
the cough peak flow generated through unassisted MI-E, manually-assisted MI-E and AFES-assisted MI-E | at end of 8 week AFES intervention
Patient's experience of using MI-E combined with AFES compared to the use of clinically established techniques | at end of 8 week AFES intervention
  Participants will be asked whether they prefer MI-E with AFES to MI-E with and without a manually assisted cough and whether they find the use of AFES more effective than the other techniques

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gollee, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Southern General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Background] Cardozo CP. Respiratory complications of spinal cord injury. J Spinal Cord Med. 2007;30(4):307-8. doi: 10.1080/10790268.2007.11753945. No abstract available. PMID 17853651
- [Background] Sancho J, Servera E, Vergara P, Marin J. Mechanical insufflation-exsufflation vs. tracheal suctioning via tracheostomy tubes for patients with amyotrophic lateral sclerosis: a pilot study. Am J Phys Med Rehabil. 2003 Oct;82(10):750-3. doi: 10.1097/01.PHM.0000087456.28979.2E. PMID 14508404
- [Background] Sivasothy P, Brown L, Smith IE, Shneerson JM. Effect of manually assisted cough and mechanical insufflation on cough flow of normal subjects, patients with chronic obstructive pulmonary disease (COPD), and patients with respiratory muscle weakness. Thorax. 2001 Jun;56(6):438-44. doi: 10.1136/thorax.56.6.438. PMID 11359958
- [Background] Bach JR. Mechanical insufflation-exsufflation. Comparison of peak expiratory flows with manually assisted and unassisted coughing techniques. Chest. 1993 Nov;104(5):1553-62. doi: 10.1378/chest.104.5.1553. PMID 8222823
- [Background] Tzeng AC, Bach JR. Prevention of pulmonary morbidity for patients with neuromuscular disease. Chest. 2000 Nov;118(5):1390-6. doi: 10.1378/chest.118.5.1390. PMID 11083691
- [Background] Linn WS, Spungen AM, Gong H Jr, Adkins RH, Bauman WA, Waters RL. Forced vital capacity in two large outpatient populations with chronic spinal cord injury. Spinal Cord. 2001 May;39(5):263-8. doi: 10.1038/sj.sc.3101155. PMID 11438842
- [Background] Bott J, Blumenthal S, Buxton M, Ellum S, Falconer C, Garrod R, Harvey A, Hughes T, Lincoln M, Mikelsons C, Potter C, Pryor J, Rimington L, Sinfield F, Thompson C, Vaughn P, White J; British Thoracic Society Physiotherapy Guideline Development Group. Guidelines for the physiotherapy management of the adult, medical, spontaneously breathing patient. Thorax. 2009 May;64 Suppl 1:i1-51. doi: 10.1136/thx.2008.110726. No abstract available. PMID 19406863
- [Background] Cheng PT, Chen CL, Wang CM, Chung CY. Effect of neuromuscular electrical stimulation on cough capacity and pulmonary function in patients with acute cervical cord injury. J Rehabil Med. 2006 Jan;38(1):32-6. doi: 10.1080/16501970510043387. PMID 16548084
- [Background] Sorli J, Kandare F, Jaeger RJ, Stanic U. Ventilatory assistance using electrical stimulation of abdominal muscles. IEEE Trans Rehabil Eng. 1996 Mar;4(1):1-6. doi: 10.1109/86.486051. PMID 8798066
- [Background] Jaeger RJ, Turba RM, Yarkony GM, Roth EJ. Cough in spinal cord injured patients: comparison of three methods to produce cough. Arch Phys Med Rehabil. 1993 Dec;74(12):1358-61. doi: 10.1016/0003-9993(93)90093-p. PMID 8018145
- [Background] Langbein WE, Maloney C, Kandare F, Stanic U, Nemchausky B, Jaeger RJ. Pulmonary function testing in spinal cord injury: effects of abdominal muscle stimulation. J Rehabil Res Dev. 2001 Sep-Oct;38(5):591-7. PMID 11732836
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882